CLINICAL TRIAL: NCT03384589
Title: A Randomized Controlled Trial to Compare a 1-dose vs. 2-dose Priming Schedule of 13-valent Pneumococcal Conjugate Vaccine in Canadian Infants; a Canadian Immunization Research Network (CIRN) Study
Brief Title: CIRN Pneumococcal Conjugate Vaccine 1 vs. 2 Dose Priming Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Immunization Research Network (Network); Alberta Children's Hospital (Other); Université de Montréal (Other); IWK Health Centre (Other); University of Calgary (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Manish Sadarangani, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H17-02645; CIRN23/CT16 (Other: UBC)
Record Dates: First submitted 2017-12-15; First posted 2017-12-27 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Invasive Pneumococcal Disease, Protection Against; Streptococcus Pneumoniae Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Intervention Model Description: Group 1: 3 doses of PCV13 (2, 4, 12 months), 2+1 Group 2: 2 doses of PCV13 (2, 12 months), 1+1
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: 3 doses of PCV13 (Active Comparator): PCV13, 0.5ml intramuscular at 2, 4 and 12 months of age
  Interventions: Biological: PCV13
- Group 2: 2 doses of PCV13 (Experimental): PCV13, 0.5ml intramuscular at 2 and 12 months of age
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: PCV13 — Vaccine against pneumococcal disease
  Other Names: Prevnar 13

SUMMARY:
This study is assessing if a reduced dosing schedule (1+1) of the 13-valent pneumococcal conjugate vaccine (PCV13) is non-inferior to the currently used schedule used in most of Canada.The vaccine is currently usually given as 3 doses at 2, 4 and 12 months of age. This study aims to find out if it is possible to achieve the same protection using just 2 doses, at 2 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant born at ≥37 weeks' gestation
* Age 2 months (+ up to 14 days) at time of first study visit
* Parent/guardian or legally authorized representative has given informed consent for their child's participation.

Exclusion Criteria:

* Already received any routine 2-month immunizations
* Previous laboratory confirmed pneumococcal disease
* Previous receipt of any pneumococcal vaccine
* Confirmed or suspected immunodeficiency, including but not limited to:

  * Congenital or acquired asplenia, or splenic dysfunction
  * B-cell (humoral), T-cell mediated, complement, or phagocytic function deficiency
  * HIV infection
  * Hematopoietic stem cell transplant (recipient)
  * Malignant neoplasms, including leukemia and lymphoma
  * Nephrotic syndrome
  * Solid organ or islet transplant (candidate or recipient)
* A family history of congenital or hereditary immunodeficiency
* Use of systemic immunosuppressive medication, including long-term corticosteroids, chemotherapy, radiation therapy, post-organ transplant therapy, intravenous immunoglobulin and/or specific monoclonal antibody therapy
* Bleeding disorder or thrombocytopenia, that contraindicates intramuscular (IM) injection and/or blood collection or taking any anti-platelet or anti-coagulant medications
* Any contraindication to vaccination as per the NACI Canadian Immunization Guide (https://www.canada.ca/en/public-health/services/canadian-immunization-guide.html, accessed 16 September 2017). Note these factors will be considered an exclusion if known at the time of trial enrollment, but specific screening and/or testing for these conditions will not be part of the trial):

  * Anaphylaxis to any vaccine or vaccine component being given during the trial, including PCV13 and other routine vaccines
  * Any other previous adverse event which in the opinion of the Investigator is a contraindication to any vaccine being given during the trial
  * Congenital malformation of the gastrointestinal tract or previous intussusception (rotavirus vaccine contraindicated)
  * Active, untreated tuberculosis (MMR, varicella, MMRV contraindicated)
* Additional factors resulting in increased risk of pneumococcal disease as per the National Advisory Committee on Immunization (NACI) Canadian Immunization Guide (16 September 2017)

  * Chronic cerebrospinal fluid (CSF) leak
  * Chronic neurologic condition that may impair clearance of oral secretions
  * Cochlear implants, including children who are due to receive implants
  * Chronic heart disease
  * Diabetes mellitus
  * Chronic kidney disease
  * Chronic liver disease, including hepatic cirrhosis due to any cause
  * Chronic lung disease
  * Sickle cell disease or other hemoglobinopathy
* Mother received pneumococcal vaccine during pregnancy
* Mother using systemic immunosuppressive medication during pregnancy, including intravenous immunoglobulin and/or specific monoclonal antibody therapy
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Temporary exclusion criteria:

- If an infant has a temperature ≥ 38°C, then vaccination (and blood and fecal sampling if due to occur at the same visit) will be postponed until resolution of fever.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of PCV13 post-booster | 13 months of age
  Serotype-specific pneumococcal IgG concentration at 1 month post-booster dose

SECONDARY OUTCOMES:
Immunogenicity of PCV13 post-priming | 5 months of age
  Serotype-specific pneumococcal IgG concentration post-priming dose(s)
Proportion of protected infants post-booster | 13 months of age
  Proportion of infants achieving serotype-specific pneumococcal IgG concentration ≥0.35 µg/ml post-booster dose
Proportion of protected infants post-priming | 5 months of age
  Proportion of infants achieving serotype-specific pneumococcal IgG concentration ≥0.35 µg/ml post-priming dose(s)
Incidence of adverse events following PCV13 | 2, 4 and 12 months of age
  Adverse events following immunization after doses of PCV13

OTHER OUTCOMES:
Storage of fecal samples for analysis of the influence of the infant microbiome on vaccine responses | 2, 4, 6 and 12 months of age
  Collection of fecal samples at time of vaccination
Immunogenicity of PCV13 after maternal pertussis immunization | 5 and 13 months
  Comparison of primary and secondary endpoints in infants born to mothers who received pertussis immunization in pregnancy vs. those that did not
Rate of nasopharyngeal colonization after vaccination with S. pneumoniae | 13 months
  Comparison of nasopharyngeal colonization rate with S. pneumoniae in Group 1 vs. Group 2

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sadarangani, MD, Principal Investigator — UBC
Locations (1):
- Vaccine Evaluation Center (University of BC at Children's Hospital), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided